CLINICAL TRIAL: NCT06080295
Title: The Involvement of the Kallikrein-Kinin System in the Pathogenesis of Postoperative Injury in Cardiac Surgery: An Observational Study
Brief Title: The Kallikrein-Kinin System in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Qin Zhang (Other)
Responsible Party: Sponsor-Investigator, Qin Zhang, phd, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20230932
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cardiosurgery
Keywords: KKS; tissue kallikrein; ;cardiosurgery;cardiopulmonary bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Preserving plasma by utilizing blood samples remaining from blood gas analysis during surgical procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We aimed to established an interlink among the kallikrein-kinin system (KKS), endothelial dysfunction and cardiac inflammation in response to cardiosurgery , using clinic investigation.

DETAILED DESCRIPTION:
The KKS, which is located on the vascular endothelium, plays a pivotal role in maintaining cardiovascular homeostasis. Tissue kallikrein (TK), a serine protease and a key enzyme of the KKS, is responsible for cleaving low-molecular-weight kininogen into bradykinin and kallidin. Under normal physiological conditions, the activation of the B2 receptor (B2R)/endothelial nitric oxide synthase (eNOS) signaling pathway leads to the transient release of nitric oxide (NO), resulting in cardiovascular protection. However, during reperfusion injury, the activation of the B1 receptor (B1R)/inducible nitric oxide synthase (iNOS) pathway leads to excessive NO production, promoting inflammation and cellular injury. Therefore, it is hypothesized that the KKS plays a critical role in the early stages of reperfusion injury during cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

1) Willing to participate in the study. 2) Age ≥ 18 years and ≤ 80 years. 3) Patients undergoing cardiac surgery: (coronary artery bypass grafting, heart valve surgery, Morrow operation, aortic dissection surgery).

Exclusion Criteria:

1) Patients with heart failure. 2) Patients experiencing adverse events during surgery. 3) Solid organ or bone marrow transplant recipients. 4) Patients with autoimmune diseases, tumors, or those who received high-dose steroid or immunosuppressant therapy within the past two months. 5) Deemed unsuitable for participation in this study by the researchers' judgment.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery: (coronary artery bypass grafting, heart valve surgery, Morrow operation, aortic dissection surgery).
Sampling Method: Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
survival | 24 hours
  survival and KKS related factors levels
Cardiac function | 24 hours
  echocardiography and Myo-cardial enzymonram
POD-postoperative delirium | 7 days
  Confusion Assessment Method for the ICU (CAM-ICU)

SECONDARY OUTCOMES:
survival | 28 days
  survival and clinical symptom

CONTACTS AND LOCATIONS:
Overall Officials: Qin Zhang, phd, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China